CLINICAL TRIAL: NCT07341672
Title: The Drug-Drug Interaction Study of Clifutinib
Brief Title: A Single-center, Randomized, Open-label, Parallel-design Clinical Study to Evaluate the Pharmacokinetic Effects of Itraconazole, Fluconazole or Efavirenz on a Single Dose of Clifutinib in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEC73543-AML-105
Record Dates: First submitted 2025-12-23; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subject
Keywords: Clifutinib
MeSH Terms: interventions — Itraconazole; Fluconazole; efavirenz

STUDY DESIGN:
Masking Description: Clifutinib,Itraconazole, Fluconazole, Efavirenz
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clifutinib (Experimental): On Day 1, subjects will receive a single dose of 40 mg Clifutinib
  Interventions: Drug: Clifutinib
- Clifutinib and Itraconazole (Active Comparator): From Day 1 to Day 49, subjects will receive Itraconazole 200mg bid, and receive single dose of 40mg Clifutinib on Day 8
  Interventions: Drug: Clifutinib; Drug: Itraconazole
- Clifutinib and Fluconazole (Active Comparator): From Day 1 to Day 49, subjects will receive Fluconazole 400mg qd, and receive single dose of 40mg Clifutinib on Day 8
  Interventions: Drug: Clifutinib; Drug: fluconazole
- Clifutinib and Efavirenz (Active Comparator): From Day 1 to Day 49, subjects will receive Efavirenz 600mg qd, and receive single dose of 40mg Clifutinib on Day 8
  Interventions: Drug: Clifutinib; Drug: efavirenz

INTERVENTIONS:
Drug: Clifutinib — The subjects are required to take Clifutinib on an empty stomach for at least 10 hours and without drinking water for 1 hour. After taking the drug, they should fast for 4 hours and refrain from drinking water for 1 hour.
Drug: Itraconazole — Itraconazole is taken orally approximately 30 minutes after the start of breakfast and lunch.
  Arms: Clifutinib and Itraconazole
Drug: fluconazole — Take fluconazole on an empty stomach
  Arms: Clifutinib and Fluconazole
Drug: efavirenz — Take efavirenz on an empty stomach
  Arms: Clifutinib and Efavirenz

SUMMARY:
Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib and the safety of the combination therapy in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consents were signed voluntarily with full understanding of the trial content, process and possible adverse reactions. Be able to complete the trial according to the requirements of the trial protocol.
2. Have no plans of fertility, sperm retrieval or egg donation during the trial, and are willing to take effective contraceptive measures within 6 months from the date of signing ICF to the end of drug administration.
3. Male or female participants aged 18 to 50 years old (including 18 and 50 years old).
4. Male participants weighed at least 50 kg and female participants weighed at least 45 kg. Body mass index (BMI) = weight (kg)/height2 (m2), with BMI in the range of 18 to 28 kg/m2 (including cutoff).

Exclusion Criteria:

1. During the screening period, physical examination, vital signs, laboratory tests(blood routine, blood biochemistry, coagulation function, urine routine), chest X-ray, abdominal ultrasound (liver, gallbladder, pancreas, spleen and kidney), ophthalmic examination and other examinations were abnormal and had clinical significance.
2. QTcF was calculated with Fridericia's correction formula QTcF = QT/RR (RR^0.33=60/ heart rate (BPM)) in patients with abnormal 12-lead electrocardiogram (ECG) or corrected QT interval (QTcF) >450 ms.
3. Any positive of hepatitis B surface antigen, hepatitis C antibody, AIDS antibody, or treponema pallidum antibody.
4. The female participants were pregnant or lactating, and the blood pregnancy results at screening and admission exceeded the upper limit of the normal value.
5. Taking any prescription medication, over-the-counter medication, any vitamin product, or herbal medicine within 14 days before screening.
6. Taking any drugs that alter liver enzyme activity, such as barbiturates, rifampicin, within 30 days before screening.
7. Taking an inhibitor or inducer of CYP3A4 within 30 days before screening.
8. Were enrolled in a clinical trial of any drug within 3 months before screening and used a trial drug, or were planning to enroll in another clinical trial during the trial.
9. Received a vaccination within 28 days before screening or planned to be vaccinated during the trial.
10. Blood donation or blood loss >450 mL within 3 months before screening; Or planned to donate blood during the trial.
11. Patients with dysphagia or a gastrointestinal, hepatic, or renal disease (whether cured or not) within 6 months before screening that can affect drug absorption or excretion.
12. Suffering from any condition that increases the risk of bleeding, such as active hemorrhoids bleeding, acute gastritis or gastric and duodenal ulcers.
13. Patients with past or present serious or chronic diseases of digestive system, urinary system, respiratory system, circulatory system, nervous system, blood system, endocrine system, immune system, mental system, etc.
14. Acute illness or concomitant medication occurred from the date of signing the informed consent to the date of first administration of the investigational drug.
15. Allergic constitution (multiple drugs and food allergy), allergic to Clifutinib or any drug component, allergic to itraconazole, fluconazole and efavirenz or any drug component.
16. The average daily smoking was more than 5 cigarettes in the 3 months before the trial, or the habitual use of nicotine-containing products, and could not quit during the trial.
17. If they had a history of alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), or were unable to abstain from alcohol during the study period, or had an alcohol breath test result greater than 0 mg per 100 mL.
18. Those with a positive urine drug screen or who had a history of drug abuse or drug use in the past 5 years.
19. Ingested chocolate, any caffeinated or xanthine-rich food or drink within 24 hours before taking the test drug, or were unable to stop taking it during the trial.
20. Had taken special diet (including dragon fruit, mango, grapefruit, etc.) or had strenuous exercise within 14 days before screening, or could not stop taking special diet or strenuous exercise during the trial; Or other factors affecting drug absorption, distribution, metabolism and excretion as judged by the researchers.
21. Those who have special requirements for diet and cannot accept a uniform diet.
22. Those who had a history of faintness in needles or blood, who had difficulty in blood collection or could not tolerate blood collection by venipuncture, or who had poor evaluation of venous blood collection.
23. Participants were deemed by the investigator to be ineligible for the trial for any reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Cmax | From Day1 to Day50
  Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib in healthy participants.
AUC0-t | From Day1 to Day50
  Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib in healthy participants.
AUC0-∞ | From Day1 to Day50
  Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib in healthy participants.
%AUCex | From Day1 to Day50
  Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib in healthy participants.
Tmax | From Day1 to Day50
  Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib in healthy participants.
t1/2 | From Day1 to Day50
  Evaluate the pharmacokinetic effects of itraconazole, fluconazole, or efavirenz on a single - dose of Clifutinib in healthy participants.

SECONDARY OUTCOMES:
Adverse event | From Day1 to Day50
  Frequency, type and severity of adverse events/serious adverse events.
ECG（Electrocardiogram） | From Day1 to Day50
  Evaluation parameters include heart rate, PR interval, QTcF and QRS interval, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Body temperature | From Day1 to Day50
  Summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Blood pressure | From Day1 to Day50
  Summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Pulse | From Day1 to Day50
  Summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No